CLINICAL TRIAL: NCT01138137
Title: Phase I Dose Escalation Study of N-acetylcysteine (NAC) Administered Intravenously (IV) in Conjunction With Intraperitoneal (IP) Administered Cisplatin and IV/IP Paclitaxel in Patients With Stage III or IV Ovarian Cancer
Brief Title: N-acetylcysteine Given IV With Cisplatin and Paclitaxel in Patients With Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding was available for the cost of the IV N-acetylcysteine (NAC).
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004229; 4229 (Other: OHSU eIRB); SOL-08005-L (Other: OHSU Knight Cancer Institute); OHSU-4229 (Other: OHSU IRB)
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Ovarian Carcinoma, Stage 3 or 4; Epithelial Ovarian Carcinoma; Primary Peritoneal Carcinoma
Keywords: ovarian cancer; epithelial ovarian cancer; peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Acetylcysteine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental)
  Interventions: Drug: Paclitaxel; Drug: N-acetylcysteine; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Dose: 135mg/m2 infused IV on Day 1 of 3 week cycle
  Dose: 60mg/m2 infused IP on Day 8 of 3 week cycle
  6 treatment cycles
Drug: N-acetylcysteine — A group of 5 subjects will be evaluated at each dose level.
  On Day 2 of each 3 week cycle, subject receives IV NAC followed by IP cisplatin.
  6 treatment cycles
  Dose escalation schema:
  Level 1: 150mg/kg
  Level 2: 300mg/kg
  Level 3: 600mg/kg
  Level 4: 800mg/kg
  Level 5: 1000mg/kg
  Level 6: 1200mg/kg
  Other Names: NAC
Drug: Cisplatin — Dose: 100mg/m2 infused IP on day 2 of each 3 week cycle 60 min after the NAC infusion
  6 treatment cycles

SUMMARY:
RATIONAL FOR STUDYING IV NAC AS POTENTIAL CHEMOPROTECTANT:

Cisplatin has shown efficacy in the treatment of subjects with epithelial ovarian cancer. Systemic toxicities associated with cisplatin include nephro, oto, and nerve toxicities. It may be possible to reduce the toxicities of cisplatin by administering it in conjunction with IV NAC. NAC may reduce cisplatin related nephro, oto, and nerve toxicities without compromising the effectiveness of the chemotherapy against the ovarian cancer cells. It is possible that this combination of drugs may in the future allow ovarian cancer patients to receive the full series of IP cisplatin-paclitaxel chemotherapy, with fewer side effects and improved survival.

It is hypothesized that the proposed treatment of stage III or IV epithelial ovarian cancer with IP cisplatin and IV/IP paclitaxel in conjunction with IV NAC will limit the neurotoxicity, nephrotoxicity and ototoxicity that is associated with cisplatin administration.

DETAILED DESCRIPTION:
OBJECTIVES:

PRIMARY:

To determine the Maximum Tolerated Dose (MTD) and assess the toxicity of IV NAC in conjunction with IP cisplatin and IV/IP paclitaxel in subjects with stage 3 or 4 epithelial ovarian cancer that has been surgically debulked

SECONDARY:

* To describe tumor response in subjects receiving treatment for previously debulked stage 3 or 4 epithelial ovarian cancer with IP cisplatin, IV/IP paclitaxel , and IV NAC.
* To describe the incidence and severity of nephrotoxicity (Creatinine Clearance (CrCl)) in subjects undergoing treatment for stage 3 or 4 epithelial ovarian cancer with IP cisplatin, IV paclitaxel and IV NAC and who have had their disease surgically debulked.
* To describe the incidence and severity of hearing loss in subjects undergoing treatment for stage 3 or 4 epithelial ovarian cancer with IP cisplatin, IV/IP paclitaxel and IV NAC and who have had their disease surgically debulked.
* To describe the incidence and severity of peripheral and autonomic neuropathy in subjects undergoing treatment for stage 3 or 4 epithelial ovarian cancer with IP cisplatin, IV/IP Taxol and IV NAC and who have had their disease surgically debulked.

OUTLINE:

Subjects will undergo chemotherapy for epithelial ovarian cancer with paclitaxel IV, 135 mg/m2 (Day 1) and IP cisplatin 100 mg/m2 (Day2), followed by Taxol IP, 60 mg/m2 (Day 8) every 3 weeks for 6 courses. Sixty minutes prior to each course of IP cisplatin, IV NAC (starting at 150 mg/kg) will be infused over 30 minutes. A dose escalation schema for NAC will be followed. Toxicity to the therapy will be graded according to the Common Terminology Criteria for Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent in accordance with institutional guidelines
* Histologically confirmed diagnosis of stage 3 or 4 epithelial ovarian or primary peritoneal carcinoma
* Have had debulking surgery with optimal tumor cytoreduction
* Standard treatment offered for ovarian cancer including systemic or intraperitoneal cisplatin with systemic taxane-based chemotherapy
* Age ≥ 18 years to ≤ 75 years
* Laboratory testing within 14 days of registration:

  * White blood cell count ≥ 2.5 x 103/mm3
  * Absolute granulocyte count ≥ 1.2 x 103/mm3
  * Platelets ≥ 100 x 103/mm3
  * Creatinine < 1.8
  * Bilirubin < 2.0
  * Serum glutamate oxaloacetate transaminase (SGOT)/Serum glutamate pyruvate transaminase (SGPT) < 2.5 x institutional upper limits of normal
* Performance status must be Eastern Cooperative Oncology Group (ECOG) < 2 (Karnofsky ≥ 50)
* Life expectancy of ≥ 60 days from the date of registration

Exclusion Criteria:

* Pregnant, positive beta human chorionic gonadotropin (hCG), or lactating
* History of clinically significant reactive airway disease
* Active significant cardiac disease as evidenced by New York Heart Association Classification for chronic heart failure (CHF), Class III or IV
* Uncontrolled (over the last 30 days) clinically significant confounding medical conditions
* Allergies or other contraindications to IP cisplatin, IV Taxol, or IV NAC.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and assess the toxicity of IV NAC | 4 years
  The MTD of IV NAC will be defined as one dose level below that which produces NCI Common Toxicity Criteria (CTC) grade 3 or 4 non-hematologic toxicity in 20% of subjects. The toxicity of NAC can be differentiated from that of the chemotherapeutic drugs as the half-life of NAC is very short and adverse effects are seen either during or very soon after the administration of NAC.

SECONDARY OUTCOMES:
To describe tumor response | 4 years
To describe the incidence and severity of nephrotoxicity | 4 years
To describe the incidence and severity of hearing loss | 4 years
To describe the incidence and severity of peripheral and autonomic neuropathy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, MD, Principal Investigator — Knight Cancer Institute at Oregon Health & Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States